CLINICAL TRIAL: NCT06968104
Title: Stimulation of the Transcutaneous Auricular Vagus Nerve for Improvement of Symptoms in Patients With Post-COVID Syndrome and ME/CFS
Brief Title: Vagus Nerve Stimulation to the Ear to Improve Symptoms in Post-COVID-19 and ME/CFS
Acronym: STIMPACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luxembourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ERP 25-024 STIMPACT
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Post-COVID / Long-COVID; ME/CFS
Keywords: Post-COVID Syndrome; ME/CFS; Fatigue; Autonomic Dysfunction; taVNS; crossover; sham condition
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic; Fatigue; Primary Dysautonomias | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: This study uses a randomized, single-blind, sham-controlled crossover design. Each participant will receive both Intervention A and Intervention B in a randomized sequence. Each intervention phase lasts 4 weeks, separated by a washout period of at least 4 weeks to reduce carryover effects. Participants will serve as their own controls, improving statistical power while minimizing between-subject variability. The study is single-blind: participants will not be informed which intervention is intended to stimulate the vagus nerve. All procedures are conducted remotely, and outcomes are assessed at multiple time points via digital tools and virtual check-ins.
Who Masked: Participant
Masking Description: This is a single-blind study. Participants are blinded to the nature of the two interventions, which are referred to as Intervention A and Intervention B. One intervention delivers active transcutaneous auricular vagus nerve stimulation (taVNS) to the cymba conchae, while the other applies stimulation to the earlobe-a site without vagal innervation-serving as a sham control. To reduce placebo and expectation effects, the sham condition is not labeled or described as such to participants. Both interventions are matched for appearance and sensation to maintain effective blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention A (Experimental): Participants in this arm will receive stimulation applied to the cymba conchae of the left ear, twice daily for 30 minutes over a 4-week period. This location is known to be innervated by the auricular branch of the vagus nerve. All participants will be trained in device use and electrode placement. Adherence will be tracked via device logs and virtual check-ins.
  Interventions: Device: transcutaneous vagus nerve stimulation
- Intervention B (Sham Comparator): Participants in this arm will receive stimulation applied to the earlobe, a site not innervated by the vagus nerve, under the same schedule: twice daily for 30 minutes over a 4-week period. The procedure, device appearance, and instructions are identical to the active condition to maintain participant blinding. Adherence is tracked identically.
  Interventions: Device: transcutaneous vagus nerve stimulation

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation — Transcutaneous auricular vagus nerve stimulation (taVNS) delivered using the CE-certified tVNS® device (tVNS Technologies GmbH). Stimulation parameters include a pulse width of 250-500 μs, frequency of 10-25 Hz, and an individually titrated intensity (typically up to 5 mA). The device operates with a 20-50% duty cycle and is used at home.
  Other Names: vagus stimulation; tVNS; taVNS
  Arms: Intervention A
Device: transcutaneous vagus nerve stimulation — Sham stimulation using the same CE-certified tVNS® device. Electrode placement is on the earlobe, which lacks vagus nerve innervation. Stimulation parameters (pulse width, frequency, intensity, duty cycle) mirror those of the active condition, with intensity adjusted to perceptual threshold to mimic the sensation of real stimulation and preserve blinding.
  Other Names: taVNS; Vagus stimulation; tVNS
  Arms: Intervention B

SUMMARY:
This study is testing whether a gentle electrical stimulation of a nerve in the ear, called the vagus nerve, can help reduce fatigue and improve symptoms in people with Post-COVID Syndrome or Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS). The treatment, known as transcutaneous auricular vagus nerve stimulation (taVNS), is non-invasive and can be done at home using a small device.

Participants will try two different types of stimulation, called Intervention A and Intervention B, to see which may be more effective. Each intervention lasts 4 weeks and will be separated by a break of at least 4 weeks.

Participants will use the device at home twice a day for 30 minutes. Fatigue, quality of life, sleep, and daily activity will be tracked through surveys and wearable devices. All parts of the study-including check-ins and data collection-will be done remotely.

The goal is to learn whether this type of at-home nerve stimulation can safely improve symptoms in people with Post-COVID Syndrome or ME/CFS.

DETAILED DESCRIPTION:
The STIMPACT study is a single-blind, randomized, controlled crossover trial designed to evaluate the efficacy of transcutaneous auricular vagus nerve stimulation (taVNS) in alleviating fatigue and autonomic dysfunction symptoms in individuals diagnosed with Post-COVID Syndrome or Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS).

Participants will undergo two distinct intervention phases, referred to as Intervention A and Intervention B, each lasting four weeks and separated by a washout period of at least four weeks to minimize potential carryover effects. The order of interventions will be randomized for each participant.

During each intervention phase, participants will self-administer 30-minute stimulation sessions twice daily using a portable device designed for home use. Adherence to the stimulation protocol will be monitored through device usage logs and regular virtual check-ins with the research team.

The primary outcome measure is the change in fatigue levels, assessed using validated instruments such as the Fatigue Severity Scale (FSS) and the Chalder Fatigue Questionnaire, alongside daily symptom tracking through electronic diaries. Secondary outcomes include assessments of quality of life (SF-36, Bell's Disability Scale), post-exertional malaise (DePaul Symptom Questionnaire - Post-Exertional Malaise subscale), autonomic function (heart rate variability metrics), sleep quality (Pittsburgh Sleep Quality Index), daytime sleepiness (Epworth Sleepiness Scale), mood (Hospital Anxiety and Depression Scale), and physical activity levels (measured via actigraphy).

Data collection will occur at baseline, mid-intervention, post-intervention, and during a follow-up period, utilizing online surveys, virtual consultations, and data synchronization from wearable devices. Statistical analyses will employ mixed-model approaches to evaluate changes in outcome measures over time and between interventions, with subgroup analyses comparing responses between the Post-COVID Syndrome and ME/CFS cohorts.

This study aims to provide robust evidence on the potential benefits of taVNS as a non-invasive, home-based therapeutic option for managing fatigue and autonomic dysfunction in these patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Post-COVID Syndrome (persistent symptoms > 3 months post-infection)
* Diagnosis of ME/CFS (following Canadian Consensus Criteria) Aged 18-65
* Moderate to severe fatigue (Fatigue Severity Scale ≥ 5)
* Stable medical regimen for at least 3 months
* Participants who are willing to follow the treatment protocol, and able to comply with remote monitoring.
* Sufficient proficiency in German or English language

Exclusion Criteria:

* Pacemaker or other implanted electronic or metallic devices
* Neurological or psychiatric disorders unrelated to ME/CFS or Post-COVID Syndrome
* Pregnancy or breastfeeding
* History of vagus nerve damage or significant ear injury
* Previous or ongoing use of taVNS
* Bradycardia (resting heart rate below 60 beats per minute)
* permanent jewelry at close proximity to the ear tragus;
* Known severe coronary disease or recent heart attack (within 5 years)
* Medications that may influence autonomic function, HRV, and fatigue

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Fatigue | From baseline to end of treatment at 4 weeks.
  Reduction in fatigue measured by the Fatigue Severity and Chalder Fatigue Scales. The FSS is a 9-item scale that measures the severity of fatigue and how much it affects the person's activities and lifestyle in patients with a variety of disorders. The items are scored on a 7 point scale with 1=strongly disagree and 7=strongly agree. The minimum score=9 and maximum score possible=63. Higher the score=greater fatigue severity. More common way of scoring: mean of all the scores with minimum score being 1 and maximum score being 7. The Chalder Fatigue Scale consists of 11 items scored on a 4-point Likert scale (0 to 3). Higher total scores reflect a greater degree of fatigue.

SECONDARY OUTCOMES:
Patient Health (Quality of life) | From baseline to end of treatment at 4 weeks.
  Improvements in quality of life, assessed by the Short Form Health Survey (SF-36). The SF-36 is a 36-item scale constructed to survey health status and quality of life (Ware & Sherbourne, 1992). Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Greater scores indicate greater functioning.
Patient Health (Ability) | From baseline to end of treatment at 4 weeks.
  Assessment of functional ability/disability using the Bell CFIDS disability scale (Bell Score). Scores from 0 to 100, lower score indicating greater disability.
Post-Exertional Malaise (PEM) | From baseline to end of treatment at 4 weeks.
  PEM measured by the DePaul Symptom Questionnaire - Post-Exertional-Malaise Subscale (DSQ-PEM)
Autonomic Function | From baseline to end of treatment at 4 weeks.
  Autonomic function evaluated through Heart Rate Variability (HRV)
Sleep Quality | From baseline to end of treatment at 4 weeks.
  Assessed by the Pittsburgh Sleep Quality Index (PSQI) and daily E-Diary entries.
Sleepiness | From baseline to end of treatment at 4 weeks.
  Measured by the Epworth Sleepiness Scale (ESS). Scores from 0 to 24:
  0-5 lower normal daytime sleepiness 6-10 normal daytime sleepiness 11-12 mild daytime symptoms 13-15 moderate daytime symptoms 16-24 severe daytime symptoms
Depression and Anxiety | From baseline to end of treatment at 4 weeks.
  Evaluated using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 questions that can be scored from 0 to 3. Seven questions relate to anxiety (indicated by an 'A') and 7 questions relate to depression (as shown by a 'D'). 0-7 = Normal; 8-10 = Borderline abnormal (borderline case); 11-21 = Abnormal (case).
Patients Activity | From baseline to end of treatment at 4 weeks.
  monitored through actigraphy (i.e. step count)

CONTACTS AND LOCATIONS:
Overall Officials: André Schulz, Prof. Dr. ; Dipl. Psych., Principal Investigator — University of Luxembourg
Locations (1):
- University of Luxembourg, Esch-sur-Alzette, Luxembourg

IPD SHARING:
Plan to Share IPD: Undecided